CLINICAL TRIAL: NCT05398419
Title: Music Interventions for the Facilitation of Sleep in the Acute Geriatric Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Collaborators: St. Mary's Hospital Foundation (Unknown)
Responsible Party: Principal Investigator, Shek Fung, Principal Investigator, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMHC-21-21
Record Dates: First submitted 2022-05-13; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Sleep Disturbance; Insomnia; Music Listening Intervention; Non-musical Sound Listening Intervention
Keywords: Sleep disturbance; Insomnia; Music; Non-musical sounds
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: It will be a 3-arm randomized controlled trial where participants will be randomized to one of the three following groups: music listening intervention involving instrumental slow tempo music, non-musical sounds involving nature sounds, or standard of care on the Geriatric Assessment Unit (control). The patients will be randomized in equal ratios to the 3 groups. Each intervention will take place over 7 consecutive nights. The music or non-musical sounds will be played throughout the whole night for each patient in those groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music group (Experimental): The participants will listen to music at bedtime and overnight for 7 consecutive nights. The music selected in our study will be pleasant instrumental slow tempo music in a major mode. It will also be low contrast (without periods of silence).
  Interventions: Other: Music listening intervention
- Non-musical sounds group (Active Comparator): The participants will listen to non-musical sounds at bedtime and overnight for 7 consecutive nights. The non-musical sounds will be low-contrast nature sounds such as waves or rain. The investigators plan to use non-musical sounds that align with the frequency range of the musical stimuli.
  Interventions: Other: Non-musical sounds listening intervention
- Standard of care (Control) (No Intervention): The participants will have no change to their usual sleep routine on the Geriatric Assessment Unit.

INTERVENTIONS:
Other: Music listening intervention — Participants will listen to the music at bedtime and overnight for 7 consecutive nights. The music will be administered via headphones (sleep headbands without a cord) that are connected via Bluetooth to an MP3 player.
  Arms: Music group
Other: Non-musical sounds listening intervention — Participants will listen to the non-musical sounds at bedtime and overnight for 7 consecutive nights. The non-musical sounds will be administered via headphones (sleep headbands without a cord) that are connected via Bluetooth to an MP3 player.
  Arms: Non-musical sounds group

SUMMARY:
Sleep disturbance is a common problem experienced by older patients, especially in the acute care setting, and has detrimental effects on patients' health and recovery. There is a keen focus on non-pharmacological interventions because of the high risk of side effects related to pharmacotherapy. Music is safe and cost-effective, and there is a growing body of evidence for its potential health benefits.

The purpose of our study is to examine the impact of music listening interventions on the facilitation of sleep for patients admitted to the geriatric assessment unit (GAU).

The investigators predict that a musical listening exercise will more effectively contribute to the facilitation of sleep compared to non-musical sounds and compared to standard of care on the GAU. The investigators plan to conduct this study as a feasibility study. It will be a 3-arm randomized controlled trial where participants will be randomized to either: (1) music listening intervention, (2) non-musical sounds involving nature sounds, or (3) standard of care on the GAU. The intervention will take place over 7 consecutive nights.

The primary outcome will be sleep quality, which will be measured objectively using sleep logs and subjectively through patients' own perspectives of their sleep through the Insomnia Severity Index. Secondary outcomes will include patients' sleep quality assessed by smart watches, which the investigators will evaluate to see if the data correlates to the sleep logs and patients' subjective view of their sleep. Other secondary outcomes will include patients' mood, level of pain, number medications used for sleep, duration of stay in hospital, patients' level of enjoyment of the music or non-musical sounds, and feasibility measures.

As this is a feasibility study, the goal is to show that it is possible to conduct a larger study with the same objectives and methodology. The ultimate goal is to create high-quality evidence to support (or refute) our hypothesis that music listening interventions are effective at facilitating sleep for patients admitted to the GAU. This would be a safe and cost-effective intervention to improve the health outcomes of this vulnerable population.

DETAILED DESCRIPTION:
Summary of background:

Sleep disturbance is a common problem experienced by older patients, especially in the acute care setting, and has detrimental effects on patients' health and recovery. There is a keen focus on non-pharmacological interventions because of the high risk of side effects related to pharmacotherapy. Music is safe and cost-effective, and there is a growing body of evidence for its potential health benefits.

Purpose:

The purpose of this study is to examine the impact of music listening interventions on the facilitation of sleep and the improvement of sleep quality for patients admitted to the geriatric assessment unit (GAU), as well as the feasibility of applying these interventions.

Hypothesis:

The investigators predict that a musical listening exercise involving instrumental slow-tempo music (STM) will more effectively contribute to the facilitation of sleep compared to non-musical sounds (nature sounds) and compared to standard of care on the GAU which involves an adapted in-hospital approach to geriatric patients.

Methods:

-Study design: The investigators plan to conduct this study as a feasibility study. It will be a 3-arm randomized controlled trial where participants will be randomized to one of the three following groups: music listening intervention involving instrumental STM, non-musical sounds involving nature sounds, or standard of care on the GAU (control). The patients will be randomized in equal ratios to the 3 groups. Each intervention will take place over 7 consecutive nights. The music or non-musical sounds will be played throughout the whole night for each patient in those groups.

The investigators note that patients' medical situation will likely change throughout their hospitalization stay and this may be a confounding factor affecting their sleep. The investigators also note that patients may be discharged prior to completing the 7-day intervention.

-Study outcomes and data collection procedure: See details in section below.

-Study population: See details in section below.

-Recruitment and consent: The investigators will provide the triage questionnaire (which contains the inclusion/exclusion criteria) to the treating physicians on the GAU at SMH to help them determine which patients would be appropriate for this study. The investigators will ask the treating physician to inform the patient that there is a research project on music and sleep and ask the patient if they would be interested in hearing more. If the patient is interested, the treating physician will then inform the research team. The research assistants will then discuss with the treating physicians regarding if the patient is able to consent to the study or not. They will then know whether to seek consent directly from the patient or from their substitute decision maker. In all cases, the research assistant will then approach the patient to explain the research project in detail and confirm the patient's eligibility and interest to participate in the study.

If the patient is deemed eligible based on the inclusion and exclusion criteria, wishes to participate in the study, and deemed capable to consent by their treating physician, the research assistant will obtain the patient's consent directly from them and provide the consent form for them to sign. If the patient's physician had deemed that the patient does not have the capacity to consent, and the patient wishes to participate in the study, the patient's substitute decision maker will be asked for consent on behalf of the patient. The consent will be done by the research assistants, not by the treating physician.

-Sample size: As this is a feasibility study, the investigators aim to enroll around 50 participants in the study, estimating that 2 patients will be enrolled every week. This sample size estimation is based on previous similar studies. A randomized controlled trial conducted in 2017 in the same patient population, specifically patients admitted to the GAU at St. Mary's Hospital, included 36 patients. This study examined the effect of music on patients' health, specifically their emotions and mobility. Furthermore, most of the studies included in two recent systematic reviews and meta-analyses examining the impact of music for the improvement of sleep quality in older patients in the community had sample sizes mostly between 40 and 60 patients.

A power calculation cannot be done as this is a feasibility study and there is too much patient heterogeneity with respect to medical and cognitive status to apply a power analysis from more homogenous study populations to the current study. The investigators plan to use the results of this study to help determine the sample size required to achieve sufficient statistical power in a subsequent larger study with the same objectives and methodology.

-Data analysis: The participants' baseline characteristics will be summarized using means and standard deviations or frequencies and percentages, as appropriate. Between-group comparisons will be performed using unpaired sample t-test, Mann-Whitney, and/or Chi-square test, as appropriate. Multiple linear or logistic regression models will be used to identify whether the interventions influenced sleep outcomes. The investigators will likely also utilize repeated-measure analysis of variance, to assess outcomes in our study.

Dissemination plan:

The investigators plan to publish a manuscript of our results in a suitable specialized journal. The results with also be presented as oral presentations at Medical Grands Rounds at St. Mary's Hospital and Geriatric Medicine Grand Rounds at the MUHC (McGill University Health Centre). Furthermore, the results will be presented at the AMGQ (Association des médecins gériatres du Québec) conference in May 2023.

Expected impact of findings:

As this is a feasibility study, the goal is to show that it is possible to conduct a larger study with the same objectives and methodology. The ultimate goal is to create high-quality evidence to support (or refute) our hypothesis that music listening interventions are effective at facilitating sleep for patients admitted to the GAU. This would be a safe and cost-effective intervention to improve the health outcomes of this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* This study will include patients admitted to the GAU at St. Mary's hospital in Montréal over the six-month study period (March to August 2022). As many of the patients admitted to the GAU have major neurocognitive disorder (MNCD), the investigators will include them in our study (MNCD of any stage, including Alzheimer's disease). Furthermore, the investigators will include patients who take medications for sleep in our study, and they will be randomized into the 3 groups like all the other participants.
* The patients' baseline characteristics will be noted upon entry into the study: admitting diagnosis, demographics (age, sex), whether they have MNCD, and their music sophistication. Patients' music sophistication will be evaluated using the General Musical Sophistication Subscale (GMSS) which is embedded within the Goldsmiths Musical Sophistication Index (Gold-MSI). Furthermore, as the investigators will be including patients who use medications for sleep in our study, the investigators will note what type of medication(s) the participants are taking. Specifically, the investigators will categorize the medications in the following categories: benzodiazepines, antidepressants, antipsychotics, melatonin or other; and the investigators will note if the indication is specifically for sleep or not.

Exclusion Criteria:

* Patients who already listen to music or non-musical sounds as part of their sleep routine.
* Patients with medical instability which limits their ability to participate in the study (determined by the patient's treating physician).
* Patients who have a diagnosis of a sleep disorder including obstructive sleep apnea and REM sleep behaviour disorder.
* Patients who are unable to communicate in English or French.
* Patients with behavioural issues that limit their participation in the study; specifically, those that have agitation or hyperactivity that limits their compliance with the intervention as can be seen in cases of severe BPSD (Behavioural and Psychological Symptoms of Dementia) or hyperactive delirium.
* Patients with severe hearing impairment, specifically those for whom their hearing impairment affects their ability to communicate their consent for this study and to listen to music.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Sleep quality measured subjectively via the Insomnia Severity Index (ISI) questionnaire | 7 days
  Sleep quality will also be measured subjectively through patients' own perspectives of their sleep with the Insomnia Severity Index (ISI) questionnaire which will be administered to the patients daily. The ISI is a questionnaire which has seven questions that pertain to participants' severity of insomnia symptoms. Participants are asked to answer each question on a scale of 0 to 4 (0 being asymptomatic and 4 being very symptomatic). The seven answers are added up to get a total score which ranges between 0 and 28. The higher the score, the more severe the insomnia is. The ISI questions will be slightly modified so that the questions focus on patients' latest night of sleep, not on their sleep over the past 2 weeks, as this questionnaire will be administered daily. The ISI has been shown to be a reliable and valid tool as an outcome measure in insomnia treatment and research in older patients.
Total sleep time measured objectively via sleep logs | 7 days
  Total sleep time will be measured objectively by sleep logs. This will be done by the overnight nurses who will complete a form in the morning where they will write down the following for each participant:
  * the time of sleep onset
  * the wake time in the morning
  * the number and duration of awakenings during the night (if there are any).
  The research assistants will pick up the form the next day to collect that data. With this information, the investigators will be able to calculate the total sleep time of each participant for each night in the study.
Number of awakenings during the night measured objectively via sleep logs | 7 days
  The number of awakenings will be measured objectively by sleep logs. This will be done by the overnight nurses who will complete a form in the morning where they will write down the number and duration of awakenings during the night (if there are any) for each participant as noted above. The research assistants will pick up the form the next day to collect that data.

SECONDARY OUTCOMES:
Total sleep time assessed via smart watches | 7 days
  The patients will wear smart watches (Samsung Galaxy Fit2) at all times throughout the study period. The smart watches assess sleep quality by tracking a set of non-staging sleep parameters including total sleep time. The data collected from the smart watches will be time stamped and extracted by the study investigator without any identifying information. The investigators will assess if the data from the smart watches correlates to patients' sleep logs and their subjective view of their sleep quality.
Sleep onset latency assessed via smart watches | 7 days
  The patients will wear smart watches (Samsung Galaxy Fit2) at all times throughout the study period. The smart watches assess sleep quality by tracking a set of non-staging sleep parameters including sleep onset latency which is defined at the time that it takes to accomplish the transition from full wakefulness to sleep.
Wake after sleep onset assessed via smart watches | 7 days
  The patients will wear smart watches (Samsung Galaxy Fit2) at all times throughout the study period. The smart watches assess sleep quality by tracking a set of non-staging sleep parameters including wake after sleep onset which refers to periods of wakefulness occurring after defined sleep onset.
Sleep efficiency assessed via smart watches | 7 days
  The patients will wear smart watches (Samsung Galaxy Fit2) at all times throughout the study period. The smart watches assess sleep quality by tracking a set of non-staging sleep parameters including sleep efficiency which is defined as the amount of time actually asleep divided by the time spent in bed.
Mood assessed via visual analog mood scale | 7 days
  The data on patients' mood will be assessed via visual analog mood scale of specifically 8 emotions: afraid, confused, sad, angry, energetic, tired, happy, and tense. The visual analog mood scale includes 8 sets of a drawing of two faces connected by a long line. A "neutral" face will appear at the top of the line and a face showing an emotion will appear at the bottom of the line. The name of the emotion the face represents will be printed beneath the face. For each emotion, the participants are asked to place a mark across the line at the point which best describes how they are feeling at that moment. The distance between the "neutral" face and the mark placed by the participant will be measured in millimeters (mm) ranging between 0 and 80 mm. The higher the distance, the more intensely the participant is feeling the associated emotion. The visual analog mood scale will be administered to the participants daily throughout the study period.
Pain level assessed via a visual analog pain scale | 7 days
  Pain level be assessed via a visual analog scale that the patients will be asked to answer daily. The visual analog pain scale is a pain scale from 0 to 10 with faces along a line, with 0 representing "no pain" and 10 representing "worst pain." Participants are asked to choose a number from 0 to 10 which best describes how they are feeling. The higher the number, the higher the level of pain.
Medications used for sleep | 7 days
  The data on the number of medications used for sleep (PRNs and regular medications) will be gathered at the nursing report in the morning after the night shift, as well as via chart review. The name of the medication, the dose, and the time of administration will be recorded.
Enjoyment of intervention | 7 days
  The investigators will assess how much the patients enjoy the selected music and non-musical sounds in our study by asking them to rate their music enjoyment on a scale of 0 to 10 and by noting their qualitative comments on the music or non-musical sounds. These questions will be asked to the patients daily.
Protocol adherence | 7 days
  Data on protocol adherence, specifically whether the patients kept their headphones on throughout the night, or whether they turned the music off (by checking the mp3 player), will be gathered at the nursing report in the morning after the night shift.
Noise level | 7 days
  The investigators plan to measure the noise level present around the participants at night by placing a sound recorder at their bedside each night.
Duration of stay in hospital | 7 days
  The data on duration of stay in hospital will be gathered via chart review.
Number of participations as a feasibility measure | 6 months
  As this is a feasibility study, the investigators will record the total number of participations in the study.
Number of refusals as a feasibility measure | 6 months
  As this is a feasibility study, the investigators will record the total number of refusals throughout the study.
Number of eligible participants as a feasibility measure | 6 months
  As this is a feasibility study, the investigators will record the total number of eligible participants throughout the study.
Number of exclusions as a feasibility measure | 6 months
  As this is a feasibility study, the investigators will record the total number of exclusions throughout the study.
Availability of the data as a feasibility measure | 6 months
  As this is a feasibility study, the investigators will record the availability of the data; more specifically, they will record how often each of the above outcome measures were not available/ not completed throughout the study.
Time needed to collect the data as a feasibility measure | 6 months
  As this is a feasibility study, the investigators will record the time needed to collect the data; more specifically, they will record the total number of 4-hour shifts that were worked by the research assistants throughout the study.
Cost of the study as a feasibility measure | 6 months
  As this is a feasibility study, the investigators will record the total cost of the study including the cost of the equipment (smart watches, headphones, MP3 players, sound recorders) and the salary of the research assistants.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Chabot, MD, MSc, Principal Investigator — McGill University
Locations (1):
- St. Mary's Hospital Center, Montreal, Quebec, Canada

DOCUMENTS (1):
  • Study Protocol (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT05398419/Prot_000.pdf